CLINICAL TRIAL: NCT02228278
Title: Text 4 Fit Project: Healthcare Text Messaging to Improve Health Outcomes and Medication Compliance in Overweight and Obese Adolescents.
Brief Title: Healthcare Text Messaging to Improve Diet, Physical Activity and Weight Loss in a Pediatric Lipid Clinic
Acronym: Text4Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400433
Record Dates: First submitted 2014-08-25; First posted 2014-08-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Obesity
Keywords: Pediatric; Obesity; Overweight; Texting; Text message; SMS; Diet; Weight Loss; Nutrition; Physical activity; BMI z-score; BMI
MeSH Terms: conditions — Pediatric Obesity; Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Group A will receive the typical clinic visits plus daily text messages
  Interventions: Behavioral: Group A
- Group B (Other): Group B will act as the control and will receive the typical clinic visits.
  Interventions: Other: Group B

INTERVENTIONS:
Behavioral: Group A — Phase 1: Group A will receive the typical clinic visits plus daily text messages for 12 weeks.
  Phase 2: Group A will receive the typical clinic visits (which includes anthropometric measures every three months, counseling on physical activity and nutrition goals by a healthcare provider and for those prescribed medication for a chronic condition, medication counseling by a healthcare provide) plus daily text messages in between visits for 3 months to support their health goals.
  Arms: Group A
Other: Group B — Phase 1: Group B will receive current standard care - clinic visits every three months anthropometric assessments and counseling on physical activity and nutrition goals by a healthcare provider, typically with no patient-provider communication between visits.
  Phase 2: Group B will initially act as the control and will receive the typical clinic visits (which includes anthropometric measures every three months, counseling on physical activity and nutrition goals by a healthcare provider, and for those prescribed medication for a chronic condition, medication counseling by a healthcare provider) with typically with no patient-provider communication between visits. After a 6-month delay, Group B will then receive the intervention which includes the typical clinic visits as stated previously plus daily text messages in between visits for 3 months to support their health goals.
  Arms: Group B

SUMMARY:
The purpose of this study is to determine if health-related text messages sent from healthcare providers to overweight and obese adolescents enrolled at a pediatric lipid clinic will result in increased adherence to their nutrition and physical activity goals and improve their weight loss. The study will also assess if the volume of texts per week impacts outcomes.

DETAILED DESCRIPTION:
Phase 1: We will recruit 5 participants the from the UF Pediatric Lipid and Obesity clinic for pre-intervention cognitive interviewing to assess acceptability of the intervention and request their input on a representative sample of text messages. Then, 20 participants will be recruited from the same clinic for the intervention (10 controls, 10 intervention participants). Controls will receive current standard care - clinic visits every three months anthropometric assessments and counseling on physical activity and nutrition goals by a healthcare provider, typically with no patient-provider communication between visits. The intervention group will receive the typical clinic visits plus daily text messages in between visits with fitness and nutrition messages to support their health goals. All participants will have anthropometric measurements at baseline, 3 and 6 months. Each participant will complete a Schwartz Diet and Activity History at 0, 3 and 6 month visits, and a post intervention survey will be completed at the 3 month time point.

Phase 2: The second phase will be a larger scale study to assess for statistically significant effects of the text messaging intervention. One hundred participants will be recruited from the UF Pediatric Lipid and Obesity Clinic, one hundred from the UF Pediatric Headache Clinic and one hundred from the Congenital Heart Center for a total of three hundred (n=300) participants at three clinic locations. Participants will be randomized at each clinic location to one of two groups, Group A (immediate intervention, n=50) or Group B (control group, delayed intervention, n=50).

Participants randomized to Group A will receive the typical clinic visits (which includes anthropometric measures every three months, counselling on physical activity and nutrition goals by a healthcare provider and for those prescribed medication for a chronic condition, medication counseling by a healthcare provide) plus daily text messages in between visits for 3 months to support their health goals. Group B will initially act as the control and will receive the typical clinic visits (which includes anthropometric measures every three months, counseling on physical activity and nutrition goals by a healthcare provider, and for those prescribed medication for a chronic condition, medication counseling by a healthcare provider) with typically with no patient-provider communication between visits. After a 6-month delay, Group B will then receive the intervention which includes the typical clinic visits as stated previously plus daily text messages in between visits for 3 months to support their health goals. Participants will be seen in clinic at standard intervals for routine follow up (typically every 3 months). Three months after participants finish receiving the text messages, the same anthropometric and medication measures (for those prescribed chronic medication) that were collected at baseline as part of routine care will be repeated. Each participant will complete a Block Food Screener and Block Physical Activity Screener at 0, 3, and 6 months. A post-intervention survey will be completed after the participants have stopped receiving text messages.

ELIGIBILITY:
Phase 1:

Inclusion Criteria:

* Adolescents age 13-17
* Overweight or obese (BMI > 85th percentile)
* Attend or will start attending UF Pediatric Lipid Clinic during the study period
* Own a cell phone that can receive text messages

Exclusion Criteria:

* Current diagnosis of a psychiatric eating disorder (anorexia nervosa or bulimia)
* Pregnancy
* Medical disease that would contraindicate moderate physical activity, as determined by clinician (MD or NP) from the Lipid Clinic

Phase 2:

Inclusion criteria

* Ages 11-21
* Overweight or obese (BMI > 85th percentile)
* Attend or will start attending UF Health Pediatric Lipid and Obesity Clinic,UF Health Pediatric Headache Clinic or UF Health Congenital Heart Center during the study period
* Own a cell phone that can receive text messages (or parent owns a cell phone that can receive text messages)

Exclusion criteria

* Current diagnosis of a psychiatric eating disorder (anorexia nervosa or bulimia)
* Pregnancy
* Medical disease that would contraindicate moderate physical activity

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability of text message intervention (Phase 1) | Change in baseline and 3 months
  This will involve a pre-study interview with a small group of subjects to assess for their opinions on the text messages and study concept. Following this, we will perform a small scale trial of the program, involving 20 participants with 10 subjects in the intervention group and 10 controls. The number of participants will most likely not be adequate to reach statistical significance in detecting differences in healthy food choices, physical activity and BMI z-score between control and experimental groups. However, this study will help guide us in establishing if this healthcare texting system functions well. In addition, it may help determine if there are any trends in improvement of the target variables that would support the need for a future, larger study.

SECONDARY OUTCOMES:
Changes from baseline proportion of healthy food choices versus unhealthy choices | Change in baseline, 3 and 6 months
  Phase 1: We aim to have our adolescent subjects fill out a Schwartz Diet and Activity History at time points 0, 3 and 6 months. We will assess their baseline food choices and then assess for changes in food habits over time, with a prediction that this text message communication will help to decrease the "negative" food choices (sugars/syrups, non whole grain starches, processed foods, sugar sweetened beverages) and increase the "positive" food (fruits/vegetables, low fat dairy, water) choices by 10% (based on screener scores pre and post intervention).
  Phase 2: Each participant will complete a Block Food Screener and Block Physical Activity Screener, instead of the Schwartz Diet and Activity History, to assess the proportion of healthy food choices versus unhealthy choices.
Changes from baseline time spent doing physical activity | Change in baseline, 3 and 6 months
  Phase 1: We aim to have our adolescent subjects complete a Schwartz Diet and Activity History at time points 0, 3 and 6 months. We will assess their baseline physical activity and then assess for changes in physical activity over time, with a prediction that this text message communication will help to decrease their sedentary time (and TV time) and increase their physical activity by 10% (based on screener scores pre and post intervention).
  Phase 2: Each participant will complete a Block Physical Activity Screener, instead of the Schwartz Diet and Activity History, to assess physical activity
Changes from baseline BMI Z-score | Change in baseline, 3 months and 6 months
  Subjects will have assessments of height, weight, age and sex at 0, 3 and 6 month clinic visits. Researchers will assess for any changes in BMI Z-score across time points.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Thompson, MD, Principal Investigator — University of Florida Health Shands Children's Hospital; Kristin A Dayton, MD, Study Director — University of Florida Shands Children's Hospital
Locations (3):
- United States (3):
  - University of Florida Gerold L Schiebler Children's Medical Services Center, Pediatric Lipid and Obesity Clinic, Gainesville, Florida
  - University of Florida Shands Medical Plaza, Pediatric Lipid and Obesity Clinic, Gainesville, Florida
  - UF Health and Congenital Heart Center, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No